CLINICAL TRIAL: NCT00156897
Title: Multicentre Double Blind Placebo Controlled Parallel Group Dose Ranging Study of ATL-962 to Assess Weight Loss, Safety and Tolerability in Obese Patients With Type II Diabetes Being Treated With Metformin, in Comparison With Orlistat
Brief Title: Efficacy and Safety of ATL-962 in Obese Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alizyme (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATL-962/175/CL
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Non-Insulin-Dependent Diabetes Mellitus; Obesity
Keywords: Non-insulin-dependent diabetes mellitus; NIDDM; Type II diabetes; Obesity; Lipase inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — cetilistat; Orlistat

INTERVENTIONS:
Drug: ATL-962
Drug: Orlistat

SUMMARY:
The purpose of this study is to investigate whether ATL-962 induces weight loss in diabetic patients and whether its safety and tolerability profile is superior to that of orlistat in such patients

DETAILED DESCRIPTION:
Obesity is a significant and increasing clinical problem. There is a need for effective therapeutic agents to help people reduce weight. ATL-962 is a lipase inhibitor which could reduce the amount of fat absorbed from a person's diet, leading to weight reduction.

In this study patients with Type II diabetes who are clinically obese will receive ATL-962 at one of three dose levels, or placebo, or orlistat (another lipase inhibitor). The study will investigate the amount of weight lost after 12 weeks' treatment and will compare the safety and tolerability profile of ATL-962 and orlistat.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* Body mass index 28-45kg/m2
* HbA1c 6%-10%

Exclusion Criteria:

* Significant weight loss in the previous 3 months
* Weight gain during the run-in period
* Other serious systemic conditions, except controlled hypertension, mild asthma, and primary hypothyroidism
* History of GI disorders
* Previous surgery for weight loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-12; Study Completion 2005-10

PRIMARY OUTCOMES:
Absolute weight loss compared to baseline

SECONDARY OUTCOMES:
Proportion of patients achieving 5% or 10% weight loss
Changes in waist circumference
Changes in lipid profiles
Changes in markers of diabetes
Incidence of gastrointestinal adverse effects
Changes in other safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kopelman, Principal Investigator — Queen Mary's School of Medicine & Dentistry, London, UK
Locations (37):
- Denmark (6):
  - Aalborg Sygehus Nord, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Hellerup
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense
- Finland (7):
  - Lääkärikeskus Minerva, Eura
  - Obesity Research Unit, Helsinki
  - Suomen Terveystalo, Jyväskylä
  - Oy Foodfiles Limited, Kuopio
  - Oulun Diakonissalaitos, Oulu
  - University of Oulu, Oulu
  - Turku University Hospital, Turku
- Netherlands (5):
  - Allevon, Den Bosch Ziekenhuis
  - Allevon, DN de Bilt
  - Zeikenhuisgroep Twente, Hengelo
  - Nederlandse Obesitas Klinik, Hilversum
  - Sint Franciscus Gasthuis, Rotterdam
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Linkoping University Hospital, Linköping
  - Karolinsaka University Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Samariterhemmets Sjukhus, Uppsala
- United Kingdom (14):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital, Bath
  - Clinical Research Centre Edgbaston, Birmingham
  - Walsgrave Hospital, Coventry
  - Glasgow Royal Infirmary, Glasgow
  - Clinical Research Centre, Crosby, Liverpool
  - Liverpool University Hospital, Liverpool
  - Queen Mary's School of Medicine & Dentistry, London
  - Hammersmith Hospital, London
  - Luton & Dunstable Hospital, Luton
  - Clinical Research Centre, Manchester
  - James Cook University Hospital, Middlesbrough
  - Royal Shrewsbury Hospital, Shrewsbury
  - Clinical Research Centre, Wigan

REFERENCES:
- [Derived] Kopelman P, Groot Gde H, Rissanen A, Rossner S, Toubro S, Palmer R, Hallam R, Bryson A, Hickling RI. Weight loss, HbA1c reduction, and tolerability of cetilistat in a randomized, placebo-controlled phase 2 trial in obese diabetics: comparison with orlistat (Xenical). Obesity (Silver Spring). 2010 Jan;18(1):108-15. doi: 10.1038/oby.2009.155. Epub 2009 May 21. PMID 19461584